CLINICAL TRIAL: NCT05740592
Title: The Influence of Different Micro-Invasive Methods on Mid-Palatal Suture Separation With Rapid Maxillary Expansion in Late Adolescence: A Randomized Clinical Trial
Brief Title: Micro-invasive Methods of Mid-palatal Sutural Separation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hayder Al Naseri, Ph.D. student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 627422
Record Dates: First submitted 2022-09-21; First posted 2023-02-23 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Maxillary Expansion
Keywords: microincision; microosteoperforation; MARPE; Hyrax; adolescents
MeSH Terms: interventions — Hyx protein, Drosophila

STUDY DESIGN:
Intervention Model Description: The first part of this study will involve a clinical trial to evaluate the efficacy of adjunctive piezoelectric sutural incision and MOPs along with maxillary expansion in terms of dentoalveolar and skeletal transverse induction in late adolescent patients.
Who Masked: Participant
Masking Description: Due to the nature of the trial, it is impossible to blind the investigator to the group once it is allocated. But the radiologist who uses CBCT will be blinded for the image capturing and thus allow for the blindness of the measurements extracted from the CBCT images that will be made at the soft tissue and skeletal and dental levels.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tooth-tooth borne RPE with MOPs (Experimental): many approaches have been established to speed up orthodontic tooth movement and to decrease adverse effects. These methods are classified as, microinvasive methods include cortectomies and distraction osteogenesis and microinvasive methods include micro-osteoperforations (MOPs) and piezocision Microtrauma to the bone showed increase the synthesis of cytokines and chemokines, which are routinely released when orthodontic forces are applied . As a result, the affected area is undergoing a faster bone regeneration process
  Interventions: Procedure: micro-osteoperforations ,microincision
- Tooth-Tooth borne RPE with Piezocision group (Experimental): Piezosurgery is an ultrasonic micro vibration-based bone cutting method. It used as a careful, promising, and soft tissue sparing method. In addition to its simplicity of use in the clinic, scientific evidence from animal models measuring wound healing and bone formation suggests that, piezosurgery has a better tissue response than traditional bone-cutting procedures
  .
  Interventions: Procedure: micro-osteoperforations ,microincision
- Tooth-Bone borne RPE group (MARPE) (Active Comparator): The MARPE is a RPE device with a rigid element that attached to palate by the aid of miniscrew, exerting the expansion force directly to the maxilla's basal bone
  Interventions: Procedure: micro-osteoperforations ,microincision

INTERVENTIONS:
Procedure: micro-osteoperforations ,microincision — Patients in MOPs group will be subjected to minimal 6 MOPs 2mm apart and corticoperforation will be conducted by using drilling bure and only 1 or 2mm bicortical in the mid-palatal suture area. Patients with the piezocision group will be subjected to minimal 3 micro incisions spaced 4mm apart and a piezoelectric device with diamond surgical tip (size: 4 mm, thickness: 0.5mm) will be used.. The MARPE technique comprises the insertion of four bicortical miniscrews adjacent to the mid-palatal suture, being two mesial and two distal to the expanding screw. Each MARPE have two arms and will be fixed to molar band by soldering.
  Other Names: hyrax

SUMMARY:
This trial aims to evaluate the effect of different micro-invasive methods (piezoelectric and micro-osteoperforation) along with tooth-tooth borne RPE compare to tooth-bone borne MARPE on the amount of mid-palatal sutural separation in late adolescent patients. Null Hypothesis There is no effect of adjunctive micro-invasive methods (piezoelectric and microosteoperforation) on mid-palatal suture separation with tooth-tooth borne RPE appliance compared to tooth-bone borne MARPE

DETAILED DESCRIPTION:
IMTD is commonly encountered in clinical practice and is treated using tooth-borne RME. Adult patients undergoing orthodontic treatment with tooth-borne RME frequently experience slight skeletal expansion, extrusion of posterior teeth, inability to open the palatal suture, and treatment relapse. Applying expansion forces directly to the midpalatal suture with bone-borne RME miniscrew implants is an alternative method. These bone-borne RME devices had more excellent orthopedic effects and fewer dentoalveolar side effects than their tooth-borne counterparts. Several factors, including the activation rate, influence the efficacy of RME residing in bone, such as the activation rate.

Clinical activation procedures for tooth-borne RME may not apply to bone-borne infections. As there is no existing consensus on standards for bone-borne RME, it is necessary to investigate expansion methods for these devices. In addition, the quality and amount of bone production rely on the rate of sutural growth, albeit to a lesser extent. A higher expansion rate has been related to increased sutural separation. However, the exact nature of this association and the most remarkable instantaneous expansion feasible without affecting sutural bone development have not been determined.

Using direct pressures with maximum instantaneous expansion to open mature midpalatal sutures can result in significant sutural stresses, and varied MTD is commonly observed clinically and controlled with tooth-borne RME. Adult patients undergoing orthodontic treatment with tooth-borne RME frequently experience slight skeletal expansion, extrusion of posterior teeth, inability to open the palatal suture, and treatment relapse. Applying expansion forces directly to the midpalatal suture with bone-borne RME miniscrew implants is an alternative method. These bone-borne RME appliances produced more robust orthopedic results and fewer dentoalveolar side effects than tooth-borne ones. Several parameters, including activation rate, influence the effectiveness ofbone-borne RME.

Clinical activation techniques for tooth-borne RME might not apply to bone-borne RME. As there is no current consensus on standards for bone-borne RME, expansion techniques for these devices require exploration. In addition, the rate of sutural expansion influences the quality and amount of bone production, albeit to a lesser extent. Although a faster expansion rate has been related to more significant sutural separation, the exact nature of this association and the most remarkable instantaneous expansion feasible without impairing sutural bone development have not been determined. Nonetheless, using direct forces with the maximal immediate expansion to open mature midpalatal sutures might result in substantial sutural strains and varying degrees of pain. SARME was utilized to assist transverse maxillary expansion in older individuals to alleviate high sutural tension and discomfort.

It has been discovered that the midpalatal suture offers the most resistance to maxillary expansion. For successful maxillary expansion in adult patients, it is necessary to overcome bone resistance at the midpalatal suture. Numerous techniques for simplifying, securing, and improving the predictability of surgical treatments for SARME, such as piezoelectric corticotomy, have been recently investigated. The latter dramatically minimises the traumatic side effects, surgical site bleeding, and procedure and healing time associated with conventional MARPE insertion techniques. During surgery, these instruments' precision enables the creation of precise, clean, and smooth geometries.

Consequently, several therapeutic applications of piezoelectric surgery in SARME and Le Fort I osteotomy and microosteoperforation with MARPE have been documented.

However, high-quality research, such as randomized clinical trials and prospective cohort studies with a well-defined appliance design and treatment protocol, is strongly encouraged to provide a higher level of evidence regarding the efficacy of rapid maxillary expansion in late-adolescent patients treated with minimally invasive techniques, such as MOPs and piezocision. However, no prior clinical trial has been conducted to examine the impact of different micro-invasive procedures on mid-palate sutural separation and rapid palatal extension in late adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the bilateral maxillary transverse deficiency.
2. Patient referred by orthodontists for SARME or MARPE.
3. Patients with developmental age in stage C or stage D maturation stages .
4. Patients without developmental deformity.
5. Good oral hygiene.
6. Patient with intact maxillary first premolars and first molars.

Exclusion Criteria:

1. Congenital maxillofacial deformities mainly cleft patients.
2. Previous orthodontic and surgical treatment on the maxilla.
3. Maxillary trauma.
4. Previous extraction in the maxillary arch.
5. Patients with periodontal disease.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-03-20 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Intraoral scanner outcomes | T0: before expansion
  the use of an intraoral scanner RW1: The arch width defines as the distance in a straight line between the palatal cusp tip of the right and left first premolars. RW2: The arch width defines as the distance in a straight line between the mesiopalatal cusp tip of the right and left first molars. PV: The palatal vault height defines as the vertical distance from the occlusal plane to the median line of the palate in the position connecting the mesiodistal center of the left and right first molars. To assess the inter and intra reliability the arch width and palatal vault height of each patient will be measured three times.
Intraoral scanner outcomes | T1:3 months after expansion
  the use of an intraoral scanner RW1: The arch width defines as the distance in a straight line between the palatal cusp tip of the right and left first premolars. RW2: The arch width defines as the distance in a straight line between the mesiopalatal cusp tip of the right and left first molars. PV: The palatal vault height defines as the vertical distance from the occlusal plane to the median line of the palate in the position connecting the mesiodistal center of the left and right first molars. To assess the inter and intra reliability the arch width and palatal vault height of each patient will be measured three times.
Intraoral scanner outcomes | T2: 6 months after expansion
  the use of an intraoral scanner RW1: The arch width defines as the distance in a straight line between the palatal cusp tip of the right and left first premolars. RW2: The arch width defines as the distance in a straight line between the mesiopalatal cusp tip of the right and left first molars. PV: The palatal vault height defines as the vertical distance from the occlusal plane to the median line of the palate in the position connecting the mesiodistal center of the left and right first molars. To assess the inter and intra reliability the arch width and palatal vault height of each patient will be measured three times.
CBCT Outcomes | T0: before expansion
  In all groups, CBCT scans will be taken before expansion , immediately after completion of the consolidation period (3month), and 6 month after placement
  NFW4: Nasal floor width measured at the area of the first premolars, 5 mm above the most inferior part of the nasal floor. NFW6: Nasal floor width measured at the area of the first molars,5 mm above the most inferior part of the nasal floor. PBW4: Palatal bone width measured at the level of a line connecting the palatal root apex of the first premolars. PBW6: Palatal bone width measured at the level of a line connecting the palatal root apex of the first molars. IRD4 (Interdental Root Distance 4): The distance between the palatal root apex of the right and left first premolars. IRD6 (Interdental Root Distance 6): The distance between the palatal root apex of the right and left first molars. ICD4 (Interdental Cusp Distance 4): The distance between the mesiopalatal cusp tip of the right and left first premolars
CBCT Outcomes | T1:3 months after expansion
  In all groups, CBCT scans will be taken before expansion , immediately after completion of the consolidation period (3month), and 6 month after placement
  NFW4: Nasal floor width measured at the area of the first premolars, 5 mm above the most inferior part of the nasal floor. NFW6: Nasal floor width measured at the area of the first molars,5 mm above the most inferior part of the nasal floor. PBW4: Palatal bone width measured at the level of a line connecting the palatal root apex of the first premolars. PBW6: Palatal bone width measured at the level of a line connecting the palatal root apex of the first molars. IRD4 (Interdental Root Distance 4): The distance between the palatal root apex of the right and left first premolars. IRD6 (Interdental Root Distance 6): The distance between the palatal root apex of the right and left first molars. ICD4 (Interdental Cusp Distance 4): The distance between the mesiopalatal cusp tip of the right and left first premolars
CBCT Outcomes | T2:6 months after expansion.
  In all groups, CBCT scans will be taken before expansion , immediately after completion of the consolidation period (3month), and 6 month after placement
  NFW4: Nasal floor width measured at the area of the first premolars, 5 mm above the most inferior part of the nasal floor. NFW6: Nasal floor width measured at the area of the first molars,5 mm above the most inferior part of the nasal floor. PBW4: Palatal bone width measured at the level of a line connecting the palatal root apex of the first premolars. PBW6: Palatal bone width measured at the level of a line connecting the palatal root apex of the first molars. IRD4 (Interdental Root Distance 4): The distance between the palatal root apex of the right and left first premolars. IRD6 (Interdental Root Distance 6): The distance between the palatal root apex of the right and left first molars. ICD4 (Interdental Cusp Distance 4): The distance between the mesiopalatal cusp tip of the right and left first premolars

SECONDARY OUTCOMES:
Treatment duration | T0: before expansion, T4:3 months after expansion, T5:6 months after expansion.
  The time from fixation to removal (time to event) will be recorded. The expansion rate, which can be calculated as the amount of expansion divided by the total number of follow-up periods for all participants, will be reported.
Treatment duration | T0: before expansion
  The time from fixation to removal (time to event) will be recorded. The expansion rate, which can be calculated as the amount of expansion divided by the total number of follow-up periods for all participants, will be reported.
Treatment duration | T1:3 months after expansion
  The time from fixation to removal (time to event) will be recorded. The expansion rate, which can be calculated as the amount of expansion divided by the total number of follow-up periods for all participants, will be reported.
Treatment duration | T2: 3 months after expansion
  The time from fixation to removal (time to event) will be recorded. The expansion rate, which can be calculated as the amount of expansion divided by the total number of follow-up periods for all participants, will be reported.
Periodontal health | T0: before expansion
  The impact of the therapy on periodontal health and supporting structures. For premolars and molars, the gingival index, probing depths, and bleeding on probing will be among the criteria, CBCT will be used to determine the extent of buccal bone resorption.
Periodontal health | T1:3 months after expansion
  The impact of the therapy on periodontal health and supporting structures. For premolars and molars, the gingival index, probing depths, and bleeding on probing will be among the criteria, CBCT will be used to determine the extent of buccal bone resorption.
Periodontal health | T2:6 months after expansion.
  The impact of the therapy on periodontal health and supporting structures. For premolars and molars, the gingival index, probing depths, and bleeding on probing will be among the criteria, CBCT will be used to determine the extent of buccal bone resorption.
Soft tissue impaction | T0: before expansion.
  Soft tissue impaction will be the third secondary outcome, which will be measured by extraoral scaner to perioral soft tissue three months following the retention period.
Soft tissue impaction | T1:3 months after expansion
  Soft tissue impaction will be the third secondary outcome, which will be measured by extraoral scaner to perioral soft tissue three months following the retention period.
Soft tissue impaction | T2:6 months after expansion.
  Soft tissue impaction will be the third secondary outcome, which will be measured by extraoral scaner to perioral soft tissue three months following the retention period.

CONTACTS AND LOCATIONS:
Overall Officials: Harraa S. Mohammed-Salih, Ph.D., Study Director — University of Baghdad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altug Atac AT, Karasu HA, Aytac D. Surgically assisted rapid maxillary expansion compared with orthopedic rapid maxillary expansion. Angle Orthod. 2006 May;76(3):353-9. doi: 10.1043/0003-3219(2006)076[0353:SARMEC]2.0.CO;2. PMID 16637711
- [Background] Baccetti T, Franchi L, McNamara JA Jr. An improved version of the cervical vertebral maturation (CVM) method for the assessment of mandibular growth. Angle Orthod. 2002 Aug;72(4):316-23. doi: 10.1043/0003-3219(2002)0722.0.CO;2. PMID 12169031